CLINICAL TRIAL: NCT02548611
Title: Intensified Loading With Prasugrel Versus Standard Loading With Clopidogrel in Invasive-treated Patients With Biomarker-Negative Angina Pectoris
Brief Title: Comparison of Loading Strategies With Antiplatelet Drugs in Patients Undergoing Elective Coronary Intervention
Acronym: SASSICAIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to low recruitment
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julinda Mehilli, Prof. Dr. med., LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE MucT002-14
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): single-dose loading with 60 mg of prasugrel pre PCI
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): loading with 600 mg of clopidogrel pre PCI
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — see arm description
  Other Names: Efient
  Arms: Prasugrel
Drug: Clopidogrel — see arm description
  Other Names: Iscover, Plavix
  Arms: Clopidogrel

SUMMARY:
Use of high loading doses of clopidogrel (antiplatelet drug) just before coronary interventions is associated with improved outcomes after coronary stenting. However the onset of platelet inhibition after clopidogrel loading takes 2 to 4 hours and its action if very variable. A way to overcome this limitation is loading with a more potent antiplatelet drug such as prasugrel. Therefore in the current study the investigators want to compare loading with 60 mg prasugrel (potent antiplatelet drug) and loading with clopidogrel (standard drug) in patients undergoing elective coronary intervention.

DETAILED DESCRIPTION:
Patients with stable or clinically unstable (biomarker-negative) angina pectoris who are in need of coronary intervention will be randomly assigned in one of the treatment strategies - 60 mg of prasugrel or 600 mg clopidogrel just prior to percutaneous coronary intervention (PCI). After PCI all patients will receive clopidogrel 75 mg/d as per standard. The patients will be monitored throughout a 30-day time frame and ischemic and bleeding events will be recorded. The study is powered to show the superiority of single-dose 60 mg prasugrel over single-dose 600 mg clopidogrel regarding the ischemic complications at 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biomarker negative stable or unstable angina pectoris
* Written informed consent
* In women with childbearing potential a pregnancy test is obligatory

Exclusion Criteria:

* Age < 18 years and >80 years
* ST-elevation MI
* Elevated cardiac biomarkers
* Subjects with known contraindications to clopidogrel treatment, which are hypersensitivity to the drug substance or any component of the product and active pathological bleeding such as peptic ulcer or intracranial hemorrhage and with known severe liver disease (Child Pugh Class C)
* Subjects with known contraindications to prasugrel treatment, which are hypersensitivity to the drug substance or any component of the product, active pathological bleeding such as peptic ulcer or intracranial hemorrhage and a history of prior transient ischemic attack (TIA) or stroke and with known severe liver disease (Child Pugh Class C)
* Chronic therapy on potent P2Y12 receptor inhibitors (ticagrelor, prasugrel)
* Pre-treatment with a loading dose of either clopidogrel, prasugrel or ticagrelor
* Simultaneous participation in another clinical trial that involves the administration of an investigational medicinal drug within 30 days prior to the start of this clinical trial
* Major surgeries in the last 6 weeks and planned surgeries within the next 6 weeks (per decision of the treating physician)
* Active bleeding
* Known or persistent abuse of medication, drugs or alcohol
* Current or planned pregnancy or nursing women, women 90 days after childbirth. Females of childbearing potential, who do not use and are not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Combined ischemic events | 30 days
  Combined outcome of all-cause death, any myocardial infarction (MI), stent thrombosis, urgent revascularization and stroke

SECONDARY OUTCOMES:
Bleeding | 30 days
  Academic Research Consortium ≥2 bleeding and TIMI classification
Peri-PCI MI Type 4a | 30 days
  according to Third Universal Definition of MI
All-cause death | 30 days
  mortality
Any myocardial infarction | 30 days
  according to SASSICAIA protocol definition
Stent thrombosis | 30 days
  according to Academic Research Consortium criteria
Urgent vessel revascularization | 30 days
  revascularization related to symptoms
cerebro-vascular events | 30 days
  stroke and TIA

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — University Hospital Munich
Locations (5):
- Germany (4):
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen, Freiburg im Breisgau, Bad Krozingen
  - Munich University Hospital, Munich, Bavaria
  - Deutsches Herzzentrum Muenchen, Munich
  - Klinikum Bogenhausen, Munich
- Heart Center Balatonfüred and Heart and Vascular Center, Balatonfüred, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehilli J, Baquet M, Hochholzer W, Mayer K, Tesche C, Aradi D, Xu Y, Thienel M, Gschwendtner S, Zadrozny M, Jochheim D, Sibbing D, Schupke S, Mansmann U, Hoffmann E, Kastrati A, Neumann FJ, Massberg S. Randomized Comparison of Intensified and Standard P2Y12-Receptor-Inhibition Before Elective Percutaneous Coronary Intervention: The SASSICAIA Trial. Circ Cardiovasc Interv. 2020 Jun;13(6):e008649. doi: 10.1161/CIRCINTERVENTIONS.119.008649. Epub 2020 Jun 12. PMID 32527192